CLINICAL TRIAL: NCT01454999
Title: Cell Phone-Based Expert Systems for Smoking Cessation
Acronym: TXT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Pacific Islands Health Care System (U.S. Federal Agency)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2009-05/PJJ 0001
Record Dates: First submitted 2011-10-14; First posted 2011-10-19 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Smoking
Keywords: veteran; smoking; stage of change; cell phone; computerized tailored intervention
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CTI (Experimental): Web-based computerized, tailored intervention (CTI) for smoking cessation, based on the transtheoretical model of change.
  Interventions: Behavioral: CTI
- CTI + text (Experimental): Web-based computerized, tailored intervention (CTI) for smoking cessation, based on the transtheoretical model of change. Tailored feedback messages based on stage of change will also be sent by cell phone.
  Interventions: Behavioral: CTI

INTERVENTIONS:
Behavioral: CTI — Web-based computerized, tailored intervention (CTI) for smoking cessation, based on the transtheoretical model of change.

SUMMARY:
This project aims to enhance the emotional and physical well-being of veterans through the reduction of smoking by utilizing a web-based, computerized tailored intervention (CTI) with feedback messages delivered via cell phone. CTIs have shown increasing promise as useful behavior change programs for improved health behaviors. A variety of modalities are to deliver personalized CTI information and feedback; however, the ubiquity and sophistication of today's wireless mobile technologies represent new modes of delivery for empirically based smoking cessation and other behavioral health interventions. The CTI is based on the empirically-supported Transtheoretical Model of Behavior Change (TTM). A web-based CTI modified for a veteran population will be used to pilot test the effectiveness of the CTI alone and CTI plus individualized text messaging enhancements. The pilot study is a randomized controlled trial to assess the cell phone's feasibility as an intervention modality for changing smoking behaviors. This will be the first study to adapt a smoking cessation Internet-based CTI to provide personalized feedback on a cell phone to reduce smoking behaviors in military veterans.

DETAILED DESCRIPTION:
Objective: This project examined the effectiveness of tailored text messages as an enhancement to a computerized tailored intervention (CTI) for smoking cessation with Veterans. It was theorized that the ubiquity and sophistication of today's wireless mobile technologies would represent new modes of delivery for empirically based smoking cessation and other behavioral health interventions. CTIs have shown increasing promise as useful behavior change programs for improved health behaviors; however, the ubiquity and sophistication of today's wireless mobile technologies represent new modes of delivery for evidence-based smoking cessation and other behavioral health interventions. The CTI was based on the Transtheoretical Model of Behavior Change (TTM) and developed by Pro-Change Behavior Systems, Inc.

Research Design: This randomized, prospective pilot employed a 2 (group) x 3 (timepoint) research design. Veteran smokers were recruited nationally from direct mailings, Facebook ads, community newsletters, posters, and flyers. In addition to the randomized control trial (RCT), a focus group (n=9) and individual usability tests (n=5) were conducted in order to assess the acceptability of the graphic user interface, questions, tailoring and program content to Veteran smokers. The pilot study tested the effectiveness of the CTI alone and CTI plus individualized text messaging enhancements in reducing smoking behavior in Veterans. In addition to smoking cessation, readiness to change other negative health behaviors � such as alcohol use, healthy eating, and exercise � was also assessed.

Summary of Research Methodology and Procedures: Usability Testing: Five separate usability tests were conducted for the CTI smoking cessation program using a combination of the Think Aloud protocol and Wizard of Oz approach. Usability testing software was used to take notes and record participant interactions with the program. Participants provided qualitative and quantitative feedback on overall presentation and usability of the program. All interview data were coded, categorized, and summarized in a feedback report so that revisions to the system could be adapted. Pilot Study: At all three timepoints, participants completed a brief Health Risk Intervention (HRI), two additional smoking assessments, and the smoking cessation (SC) intervention. The HRI assessment determined baseline readiness to change for smoking and several other related health behaviors, and the smoking cessation intervention provided assessment and feedback about participants' confidence to quit smoking, decisional balance, and use of various change strategies. Following the baseline HRI and SC intervention, the CTI system randomized participants into either the treatment group (Tx), who also received the CTI only, or the treatment-plus group (Tx-plus), who received the CTI and tailored text messages. The study was conducted as entirely anonymous. All participants were given three months' access to the web-based CTI system. The Tx participants received only the online feedback narratives/report that all participants received upon completion of the online Smoking Cessation intervention. Tx-plus participants also received individualized text messages on their cell phones 2-5 times per week (the number of messages correlated with the participant's stage of change) that provide expert guidance, encouragement, and reminders that support their smoking cessation efforts.

Findings: Four-hundred and forty-six Veterans were recruited at baseline. All participants were active smokers, distributed across the stages of change as 11.9% in Precontemplation (n=53; not intending to change in the next 6 months); 63% in Contemplation (n=281; intending to change in the next 6 months), and 25.1% in Preparation (n=112; intending to change in the next 30 days). Two-hundred and thirty-five individuals (52.7%) completed the one-month and three-month follow-ups: n=116 in the treatment group (CTI only; Tx) and n=119 in the treatment-plus group (CTI plus text messages; Tx-plus). Results indicated that the CTI-plus-text-messaging intervention outperformed the CTI-only intervention at an unprecedented quit rate. For those participants in the Tx group 32.8% had quit smoking at three-month follow-up; however, those in the Tx-plus group had quit rates of 43.2%. These findings are highly encouraging, and exceed those quit rates found for other CTI interventions for both groups by almost 15% (Krebs, Prochaska & Rossi, 2010).

Summary of Participant Experiences: While data are available only for those participants who completed the study, indications from the User Satisfaction Scale, as well as the open-ended questions, were that Veterans found the CTI and tailored text messages to be both appropriate and relevant. In addition, participants in the Tx-plus group also indicated that the text messages were helpful, timely and useful. There were no adverse events to report.

Summary of Current Risk - Potential Benefit Assessment based on Study Results: This study was able to demonstrate that the TTM is an appropriate model to promote multiple behavior change in Veterans. Furthermore, the addition of tailored text messages increased the effect of the smoking cessation intervention (CTI) and improved quit rates in the Tx-plus group to levels that are unprecedented in the literature. Additionally, individuals who were at risk for other health behaviors progressed to A or M without intervention. For Veterans who are not ready for in-person psychotherapy, have practical issues attending therapy sessions, or fear stigma associated with seeking mental health care, this Veteran-tailored, motivational enhancement CTI may provide unique benefits. In addition, Veterans who smoke and have comorbid behavioral risk factors may find this CTI sufficient to resolve their problems. In this sense, the adapted CTI will make evidence-based mental health care more accessible to Veterans in need without adding concerns about stigma and costs.

Impact/Significance: This is the Final Abstract for this research project. This study was the first to adapt a smoking cessation Internet-based CTI to provide personalized feedback on a cell phone to reduce smoking behaviors in military Veterans. The findings suggest that behavior change interventions can be successfully delivered to Veterans via the Internet, and that tailored text messaging can significantly enhance the intervention effects.

ELIGIBILITY:
Inclusion Criteria:

Male and female veterans, OIF/OEF service preferred 18 years or older Current cigarette smoker Own cell phone with text messaging capabilities Ability to read and comprehend English Beginner level computer literacy Access to a computer with Internet connectivity

Exclusion Criteria:

Lack of basic computer literacy Non-smoker (includes smokeless tobacco use) Unable to read and comprehend English No access to computer with Internet connectivity (applicable if no project computer with Internet access can be arranged) Non-owner of cell phone with text messaging capabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2009-09; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Smoking prevalence | 3-months
  7-day point prevalence (self-report)

SECONDARY OUTCOMES:
Stage of Change | 3 months
  Progress through states of change for smoking cessation

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J Jordan, PhD, Principal Investigator — Pacific Health Research & Education Institute
Locations (1):
- VA Pacific Islands Health Care System, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No